CLINICAL TRIAL: NCT06643091
Title: Nintedanib Treatment in Unicentric Castleman Disease
Acronym: NUCastle
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP230820
Record Dates: First submitted 2024-09-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Castleman Disease
Keywords: Castleman disease
MeSH Terms: conditions — Castleman Disease | interventions — nintedanib

STUDY DESIGN:
Intervention Model Description: Multicenter open label and single-arm phase II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients aged 18 and over with unicentric hyalino-vascular Castleman's disease (Experimental)
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Nintedanib150 mg twice a day for 6 months Or Nintedanib 100mg twice a day in case of dose adjustment Oral route (during meals)

SUMMARY:
Unicentric Castleman Disease (UCD) is a rare non-malignant localised disease involving one or more lymph nodes, associating germinal centre atrophy, mantle zone thickening and intense vascular proliferation penetrating the germinal centres. Patients usually seek medical attention because of a localised, sometimes compressive, lymph node or the development of life-threatening autoimmune complications (paraneoplastic pemphigus or PNP or myasthenia gravis or MG). The best treatment option is complete surgical excision, but it has been recently demonstrated that up to half of the patients cannot undergo surgery. In these patients, an efficient medical approach needs be defined, as no current medical treatment has demonstrated to lower morbidity and mortality. The cause of UCD is currently unknown and current data favour a scenario of stromal impairment leading to the loss of lymph node architecture rather than one of a primary hematopoietic disease. UCD lesions are often associated with synchronous follicular dendritic cell (FDC) proliferation and can sometimes evolve towards a true FDC sarcoma (FDCS), indicating a possible role for FDC, a germinal centre stromal cell component, in UCD pathogenesis. A recurrent somatic activating mutation in PDGFRB (p.N666S) has been recently described in the CD45 negative (non-hematopoietic) compartment of up to 17% UCD specimens. Moreover, activation of the VEGFR pathway is thought to play a role in the development of the disease, especially in the increased vascularity characteristic of the UCD lesion.

Nintedanib is a commercially available tyrosine-kinase inhibitor targeting PDGF, VEGF and FGF receptors. The drug has obtained European Market Authorization in 2015 for the treatment of Non-Small Cell Lung Cancer and Idiopathic Pulmonary Fibrosis with a satisfactory safety profile. The hypothesis is that nintedanib could benefit patients with unresectable or partially resectable UCD.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ (equal to or greater than) 18 years
2. Written informed consent
3. Biopsy-proven diagnosis of hyaline-vascular Unicentric Castleman disease
4. Unresectable or partially resectable UCD lesion or surgery refusal
5. Available oral route
6. Affiliated to National French social security system (registered or being a beneficiary of such a scheme)
7. Women of childbearing potential should be advised and agree to avoid becoming pregnant while receiving treatment and to use highly effective contraceptive methods at initiation of, during and at least 3 months after the last dose of treatment; pregnancy testing must be conducted prior to treatment and during treatment as appropriate; breast-feeding should be discontinued during treatment
8. In male patients, with WOCBP partner(s), willingness to use adequate contraceptive measures to prevent his partner from becoming pregnant during the study, prior to administration of the first dose of study treatment until 3 months after the last dose of study treatment

Exclusion Criteria:

1. Synchronous Follicular Dendritic Cell sarcoma
2. Known hypersensitivity to nintedanib, soy or peanut or to any of the excipients of the experimental drug, or known hypersensitivity to the auxiliary drugs listed or to any of their excipients.
3. For women of childbearing age: negative serum or urine pregnancy test at inclusion and confirmed each month during the study, up to 3 months after the last dose.
4. Inability to obtain informed consent
5. Patients under legal protection
6. Liver transaminases (AST and/or ALT) >3N
7. End-stage liver disease (Child B or C cirrhosis)
8. End-stage renal failure (CrCl<30 mL/min)
9. Severe hemorrhagic or thromboembolic events in the past 6 months
10. Uncontrolled systemic illness such as chronic heart failure, unstable angina, hypertension; history of myocardial infarction or stroke or aneurysm
11. Major injuries in the 10 days prior to start of the study, or Recent surgery with inadequate wound healing, or Abdominal surgery in the past 4 weeks.
12. Severe pulmonary hypertension
13. Bleeding risk, any of the following:

    1. Known genetic predisposition to bleeding.
    2. Patients who require

1. Fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, direct thrombin inhibitors, heparin, hirudin) 2. High dose antiplatelet therapy corresponding to a combination of two anti-platelet aggregation treatment (aspirin + an Inhibitor of P2Y12 receptor) 14. Contraindication to the experimental drug or auxiliary drugs listed 15. Patients under guardianship or curatorship and protected adults or unable to consent 16. Enrollment in another interventional study (ongoing at the time of inclusion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Best response | Up to 6 months
  Best response over 6 months defined as >30% decrease from baseline in Total Lesion Glycolysis (TLG) measured by 18F FDG PET/CT performed at M3 and M6

SECONDARY OUTCOMES:
Number of adverse events | Up to 9 months
Number of serious adverse events | Up to 9 months
Nindetanib discontinuation | Up to 9 months
Size of the lesion | At 3 months
  Variation from baseline
Ssize of the lesion | At 6 months
  Variation from baseline
Variation from baseline in Standardized Uptake Value of the lesion | At 3 months
Variation from baseline in Standardized Uptake Value of the lesion | At 6 months
Variation from baseline in Total Lesion Glycolysis (TLG) percentage of the lesion | At 3 months
Variation from baseline in Total Lesion Glycolysis (TLG) percentage of the lesion | At 6 months
Change in the status of non-resectability of the Unicentric Castleman Disease lesion | At 6 months
Pemphigus disease area index (for Paraneoplastic pemphigus) | At 1 month
  Evolution of autoimmune-related complications by a score developped by the International Pemphigus Definitions Committee. It evaluates 3 components : skin, scalp, and mucous membranes assessing for each one activity and damage. The score varies between 0 to 263, the higher the score, he more severe the disease.
Pemphigus disease area index (for Paraneoplastic pemphigus) | At 3 months
  Evolution of autoimmune-related complications by a score developped by the International Pemphigus Definitions Committee. It evaluates 3 components : skin, scalp, and mucous membranes assessing for each one activity and damage. The score varies between 0 to 263, the higher the score, he more severe the disease.
Pemphigus disease area index (for Paraneoplastic pemphigus) | At 9 months
  Evolution of autoimmune-related complications by a score developped by the International Pemphigus Definitions Committee. It evaluates 3 components : skin, scalp, and mucous membranes assessing for each one activity and damage. The score varies between 0 to 263, the higher the score, he more severe the disease.
For bronchiolitis obliterans : change from baseline of the percent of predicted forced expiratory volume in 1 second (FEV1) | At 3 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline of the percent of predicted forced expiratory volume in 1 second (FEV1) | At 6 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline of the percent of predicted forced expiratory volume in 1 second (FEV1) | At 9 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline in forced vital capacityin forced vital capacity | At 3 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline in forced vital capacityin forced vital capacity | At 6 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline in forced vital capacityin forced vital capacity | At 9 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline in total lung capacity | At 3 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline in total lung capacity | At 6 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline in total lung capacity | At 9 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline in Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) | At 3 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline in Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) | At 6 months
  Evolution of autoimmune-related complications
For bronchiolitis obliterans : change from baseline in Diffusing Capacity of the Lung for Carbon Monoxide (DLCO) | At 9 months
  Evolution of autoimmune-related complications
For Paraneoplastic pemphigus/Bronchiolitis Obliterans: serum antibody titers | At 3 months
  anti desmoglein 1/3, anti desmoplakin, anti envoplakin, anti periplakin
For Paraneoplastic pemphigus/Bronchiolitis Obliterans: serum antibody titers | At 6 months
  anti desmoglein 1/3, anti desmoplakin, anti envoplakin, anti periplakin
For Paraneoplastic pemphigus/Bronchiolitis Obliterans: serum antibody titers | At 9 months
  anti desmoglein 1/3, anti desmoplakin, anti envoplakin, anti periplakin
For Myasthenia gravis : change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) profile score | At 1 month
  8 items score ranging from 0 (normal) to 24 (most severe).
For Myasthenia gravis : change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) profile score | At 3 months
  8 items score ranging from 0 (normal) to 24 (most severe).
For Myasthenia gravis : change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) profile score | At 6 months
  8 items score ranging from 0 (normal) to 24 (most severe).
For Myasthenia gravis : change from baseline in Myasthenia Gravis Activities of Daily Living (MG-ADL) profile score | At 9 months
  8 items score ranging from 0 (normal) to 24 (most severe).
For Myasthenia gravis : anti AchR/MusK titers | At 3 months
For Myasthenia gravis : anti AchR/MusK titers | At 6 months
For Myasthenia gravis : anti AchR/MusK titers | At 9 months
Evaluation of the mutational status of PDGFRB (Platelet Derived Growth Factor Receptor B) of the lesion and correlation with treatment response | At 3 months
  Treatment response is evaluated by variation in size, SUV (Standardized Uptake Value), TLG (Total Lesion Glycolysis)
Evaluation of the mutational status of PDGFRB (Platelet Derived Growth Factor Receptor B) of the lesion and correlation with treatment response | At 6 months
  Treatment response is evaluated by variation in size, SUV (Standardized Uptake Value) , TLG (Total Lesion Glycolysis)
Nintedanib residual plasma concentration | At 1 month
Nintedanib residual plasma concentration | At 3 months
Nintedanib residual plasma concentration | At 6 months

IPD SHARING:
Plan to Share IPD: Undecided